CLINICAL TRIAL: NCT02327247
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single-dose, Crossover, Bioequivalence Study Comparing Felodipine Extended Release Tablet (Containing Felodipine 10 mg) of OHM Laboratories Inc (A Subsidiary of Ranbaxy Pharmaceuticals Inc) With PLENDIL® Extended Release Tablet (Containing Felodipine 10 mg) Manufactured by Merck & Co. Inc. for AstraZeneca in Healthy, Adult, Male, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Felodipine ER Tablets 10 mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 243_FELOD_08
Record Dates: First submitted 2014-12-04; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Felodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Felodipine Extended Release Tablets USP 10 mg
  Interventions: Drug: Felodipine
- Reference (Active Comparator): Plendil® Extended release tablets 10 mg
  Interventions: Drug: PLENDIL®

INTERVENTIONS:
Drug: Felodipine — Extended Release Tablets, 10mg
  Arms: Test
Drug: PLENDIL® — Extended Release Tablets, 10mg
  Arms: Reference

SUMMARY:
The study was conducted as an open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioequivalence study comparing Felodipine extended release tablets USP 10 mg (containing felodipine 10 mg) manufactured by OHM Laboratories, Inc., NJ, 08901 with PLENDIL® extended release tablets 10 mg (containing felodipine 10 mg) manufactured by Merck & Co. Inc. Whitehouse Station, NJ 08889 USA for AstraZeneca LP Wilmington, DE 19850 in healthy, adult, male, human subjects under fasting condition.

DETAILED DESCRIPTION:
All the subjects were subjected to breath test for alcohol and test for drugs of abuse (opioids and cannabinoids) prior to admission in each period. Only subjects with negative results in these tests were preceded for further activities.

Following an overnight fast of at least 10 hour, a single oral dose of felodipine extended release tablet (containing felodipine 10 mg) of either test or reference formulation was administered during each period of the study, along with 240 mL of drinking water at ambient temperature under low light condition .

During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis) at baseline. Adverse event monitoring was done throughout the study. Laboratory parameters of hematology and biochemistry (except blood glucose and cholesterol) were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Volunteers who met the following criteria were included in the study

* Were in the age range of 18-45 years
* Were neither overweight nor underweight for their height as per the Life Insurance Corporation of India height/weight chart for non-medical cases
* Had voluntarily given written informed consent to participate in this study
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study

Exclusion Criteria:

* History of known hypersensitivity to Felodipine, related drugs and or any other drug
* Individuals with systolic blood pressure <100 mmHg or >140mmHg diastolic blood pressure < 60 mmHg or >90 mmHg, at the time of admission in period I
* History of chronic headache, dizziness and syncope
* History of peripheral edema
* History of grapefruit juice and / or grapefruit supplements intake in past 48 hours
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations
* Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection
* Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for hemoglobin, total white blood cells count, differential WBC count or platelet count
* Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive)
* Clinically abnormal ECG or Chest X-ray
* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma head-injury or coma
* History of any psychiatric illness which might impair the ability to provide written informed consent
* Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period
* Use of any enzyme modifying drugs within 30 days prior to Day 1 of the study
* Participation in any clinical trial within 12 weeks preceding Day 1 of the study
* Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in the past 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) aof Felodipine | 0-72 hrs
Peak Plasma Concentration (Cmax) of Felodipine | 0-72 hrs

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm